CLINICAL TRIAL: NCT00300768
Title: A Randomized, Single-Ascending Dose, Ivermectin-Controlled, Double-Blind, Safety, Tolerability, Pharmacokinetic, and Efficacy Study Of Orally Administered Moxidectin In Subjects With Onchocerca Volvulus Infection
Brief Title: Study Evaluating Orally Administered Moxidectin In Subjects With Onchocerca Volvulus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3110A1-200-GH; B1751004 (Other: Protocol ID: Pfizer); OCRC 33 (Other: Protocol ID: WHO, OCRC)
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-11

CONDITIONS: Onchocerciasis
Keywords: onchocerciasis; onchocerca volvulus; river blindness; ivermectin; moxidectin
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — moxidectin; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 2 mg moxidectin (Experimental): 2 mg moxidectin (Dose-escalation 1st step)
  Interventions: Drug: 2 mg moxidectin
- Ivermectin 150 mcg/kg (Active Comparator): Active comparator arm (ivermectin 150 mcg/kg).
  Interventions: Drug: ivermectin 150 mcg/kg
- 4 mg moxidectin (Experimental): 4 mg moxidectin (dose escalation second step)
  Interventions: Drug: 4 mg moxidectin
- 8 mg moxidectin (Experimental): 8 mg moxidectin (dose escalation third step)
  Interventions: Drug: 8 mg moxidectin

INTERVENTIONS:
Drug: 2 mg moxidectin — Single-dose, tablet encapsulated for blinding
  Arms: 2 mg moxidectin
Drug: ivermectin 150 mcg/kg — Single-dose, tablets encapsulated for blinding
  Arms: Ivermectin 150 mcg/kg
Drug: 4 mg moxidectin — Single dose, tablets encapsulated for blinding
  Arms: 4 mg moxidectin
Drug: 8 mg moxidectin — single dose, tablets encapsulated for blinding
  Arms: 8 mg moxidectin

SUMMARY:
The primary purpose of this study was to determine the safety and tolerability of moxidectin in subjects infected with Onchocerca volvulus (a parasitic worm).

DETAILED DESCRIPTION:
This was a phase 2, randomized, ivermectin-controlled, double-blind, single-ascending-dose, parallel design, inpatient/outpatient study of moxidectin administered to subjects of both sexes with different degrees of severity of O. volvulus infection. The study was conducted at a single site in Ghana.

Secondary objects are to determine the pharmacokinetics of moxidectin, to obtain initial indication of the efficacy in terms of long term effect on skin microfilaria levels and an indication of the effect on the macrofilaria that may underlie the effect on skin microfilaria levels.

Subjects were enrolled in consecutive cohorts to receive a single oral dose of 2 mg, 4 mg or 8 mg or moxidectin or ivermectin 150 µg/kg by severity of infection, based on the mean of the skin microfilariae densities at each of 4 body locations, both iliac crests and calves.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed (or thumb-printed), and dated informed consent
2. Aged 18 to 60 years, inclusive
3. Body weight ≥ 40 kg for women and ≥ 45 kg for men
4. Nonpregnant, nonbreastfeeding women. Women of child bearing potential must agree to use birth control during the first 150 days after treatment.
5. Healthy, as determined by a physician on the basis of a physical examination, ECG, and a thorough review of the medical history and clinical laboratory results
6. Adequate hematologic, renal, and hepatic function
7. Skin microfilarial density within the required range for the cohort

Exclusion Criteria:

1. Participation in any studies other than purely observational ones, within 4 weeks before test article administration.
2. Any vaccination within 4 weeks before test article administration
3. Acute infection requiring therapy within the last 10 days before test article administration
4. Administration of any medication (with the exception of medication required to treat any reactions during the screening fluorescein angiography (chlorpheniramine) or paracetamol) or herbal preparation within 10 days prior to test article administration or any condition currently requiring regular medication
5. Clinically significant ECG abnormalities or history of cardiac abnormality
6. Past or current history of neurological or neuropsychiatric disease or epilepsy
7. Subjects with orthostatic hypotension at the screening evaluation
8. History of drug or alcohol abuse or regular use of ≥ 3 cigarettes per day
9. Use of alcohol or other drugs of abuse within 72 hours before test article administration
10. Any condition, in the investigator's opinion, that places the subject at undue risk
11. Subjects who have donated blood within 8 weeks before study entry
12. Subjects with ocular onchocerciasis in cohorts intended to enroll subjects with mild infection. Ocular onchocerciasis is defined by the presence of live or dead microfilariae, onchocercal punctate opacities, onchocercal lesions of the posterior segment or lesions that mimic those seen in onchocerciasis.
13. Subjects with hyperreactive onchodermatitis
14. Antifilarial therapy within the previous 5 years
15. Coincidental infection with Loa Loa
16. Female subjects of childbearing potential with a contraindication to DMPA if not on Norplant
17. Any other condition which the investigator feels would exclude the subject from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2006-09-06 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11-29 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical adverse events and clinically significant laboratory test results | Duration of follow up (18 months)

SECONDARY OUTCOMES:
Skin mf counts at day 8 and months 1, 2, 3, 6, 12 and 18 | day 8 and months 1, 2, 3, 6, 12, 18
Nodulectomy at 18 months | 18 months
Pharmacokinetics (PKs) at days 1, 2, 4, 13, and 18 and months 1, 2, 3, 6 and 12 | days 1, 2, 4, 13, and 18 and months 1, 2, 3, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Opoku, MD, Principal Investigator — Onchocerciasis Chemotherapy Research Center, Hohoe, Ghana
Locations (1):
- Onchocerciasis Chemotherapy Research Center, Hohoe, Volta Region, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Awadzi K, Opoku NO, Attah SK, Lazdins-Helds J, Kuesel AC. A randomized, single-ascending-dose, ivermectin-controlled, double-blind study of moxidectin in Onchocerca volvulus infection. PLoS Negl Trop Dis. 2014 Jun 26;8(6):e2953. doi: 10.1371/journal.pntd.0002953. eCollection 2014 Jun. PMID 24968000
- See also: Awadzi et al 2014 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4072596/pdf/pntd.0002953.pdf